CLINICAL TRIAL: NCT06010043
Title: "Dumpling Suture Method" Versus Traditional Suture Method of Protective Loop Ileostomy in Laparoscopic Anterior Rectal Resection With Specimen Extraction Via Stoma: a Retrospective Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Tingyu Wu, Principal Investigator, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: XHEC-2023-D-146
Record Dates: First submitted 2023-08-21; First posted 2023-08-24 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Ileostomy; Complications
Keywords: ileostomy; complications; NOSES; stoma suture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Dumpling suture" for ileostomy (Experimental): The stoma is fixed with sutures in a skin fold method, and the incision is progressively reduced in a process similar to the process of folding and pinching the Chinese small dumplings. This procedure may reduce stoma complications by progressively reducing the incision and realizing the effect of hiding the skin incision.
  Interventions: Procedure: Suturing of ileostomy using "Dumpling suture method"
- Traditional suture for ileostomy (Other): The stoma was fixed at the skin using traditional sutures. The incision is narrowed by 2-3 interrupted sutures at the distal and proximal ends of the skin incision on the abdominal wall. The stoma is then fixed at the right lower abdominal incision with sutures.
  Interventions: Procedure: Suturing of ileostomy using Traditional suture method

INTERVENTIONS:
Procedure: Suturing of ileostomy using "Dumpling suture method" — Suturing of ileostomy using "Dumpling suture method"
  Arms: "Dumpling suture" for ileostomy
Procedure: Suturing of ileostomy using Traditional suture method — Suturing of ileostomy using Traditional suture method
  Arms: Traditional suture for ileostomy

SUMMARY:
Natural Orifice Specimen Extraction Surgery (NOSES), which involves obtaining specimens from the abdominal cavity without any incisions, has attracted much attention in recent years, and it has been widely popularized in the treatment of rectal cancer because of its postoperative non-incision, advantages of less trauma, quicker recovery, and postoperative aesthetics. Anastomotic fistula is a serious complication of rectal cancer surgery. For patients at high risk of anastomotic fistula, prophylactic ileostomy is often performed intraoperatively to divert feces and protect the anastomosis. For such patients, rectal anterior resection surgery with specimen extraction via stoma (NOSES with specimen extraction via stoma) is usually performed, borrowing a prophylactic stoma incision to retrieve the specimen, and also realizing the absence of additional abdominal incision. However, this procedure is prone to stoma infection and has a high complication rate (20-40%), which limits the popularization of NOSES surgery and is an urgent clinical problem. Our center has proposed a new stoma closure method (Dumpling Suture Method), which reduces the size of the incision by folding the suture to achieve the effect of hiding the skin incision and reduce stoma infection. The study aimed to introduce the "Dumpling suture method" of protective loop ileostomy in laparoscopic anterior resection and compare this new method with the traditional method. From August 1st 2019 to August 1st 2023, 22 cases of the new procedure were completed in our center, and 30 patients with stoma closure by the traditional method were included in the same period for control purposes. A retrospective analysis was conducted on 52 patients in the study center, and the intraoperative details and postoperative outcomes of the two groups were measured.

ELIGIBILITY:
Inclusion Criteria:

1. All patients underwent successful laparoscopic anterior rectal resection plus protective loop ileostomy with specimen extraction through stoma incision;
2. All patients were pathologically diagnosed with rectal carcinoma or ulcerative colitis;
3. Patients aged 18 - 80 years
4. ASA (American Society of Anesthesiologists) classification ≤ grade 3.
5. Patient participate voluntarily and sign an informed consent form

Exclusion Criteria:

1. Patients with distant metastasis;
2. Patients with colon cancer;
3. Patients with a history of previous abdominal surgery;
4. ASA (American Society of Anesthesiologists) classification > grade 3;
5. Patients who underwent emergency surgery;
6. Patients who underwent surgery ≤ 3 weeks from the last chemotherapy ;
7. Patients lost to follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Complication rate of stoma | Day 30 after surgery
  Observe and assess for stoma complications

SECONDARY OUTCOMES:
Stoma DET（Discoloration，Erosion and Tissue overgrowth） score | Day 30 after surgery
  Measure the state of the skin around the stoma and the corresponding lesion area, ranging from 0-15, higher scores mean a worse outcome of stoma
Stoma Pain Score | Day 30 after surgery
  Measurement of stoma pain level using numerical rating scale，ranging from 0-10, higher scores mean a worse outcome of pain
Quality of life scale score for patients with stoma | Day 30 after surgery
  Measurement of quality of life for patients with stoma using City of Hope Quality of Life-Ostomy Questionnaire (CHO-QOL-OQ), ranging from 0-3200, higher scores mean a worse outcome of quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
In this study personal information and data such as patient history, physical examination results, surgical records, and study questionnaire data will be collected. These data will be used to evaluate the efficacy and safety of the new procedure and for academic publication. The researcher will treat the patients' personal data confidentially and anonymize the data and information in any public release of the results of the study.
Supporting Information: Study Protocol, SAP, CSR